CLINICAL TRIAL: NCT02780570
Title: Small Volume Plasma Exchange (SVPE) for Guillain-Barré Syndrome Patients in Bangladesh: A Safety and Feasibility Study
Brief Title: Small Volume Plasma Exchange (SVPE) for Guillain-Barré Syndrome (GBS) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: GBS-CIDP Foundation International (Unknown); National Institute of Neurosciences and Hospital, Dhaka (Other Government); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-15086
Record Dates: First submitted 2016-04-10; First posted 2016-05-23 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Guillain-Barré Syndrome
Keywords: SVPE; intravenous immunoglobulin; plasmapheresis
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GBS patients (Active Comparator): Small Volume Plasma Exchange
  Interventions: Procedure: Small Volume Plasma Exchange
- non-GBS (No Intervention): non-GBS patients with central venous catheter

INTERVENTIONS:
Procedure: Small Volume Plasma Exchange — Six sessions will be done daily for consecutive 8 days (total 48 sessions). 7 ml/body weight blood will be drawn at each session and will be separated into plasma and blood cells. Blood cells will be infused back to the patients and plasma will replaced by equal volume of fresh frozen plasma and colloid solution. At the end of each day 1200 ml plasma (total 9600 ml in 48 sessions) will be removed.
  Arms: GBS patients

SUMMARY:
Guillain-Barré syndrome (GBS) is the commonest form of acute flaccid paralysis and the incidence is high in low-income countries. In Bangladesh, most GBS patients are poor. Therefore patients cannot afford expensive specific treatments like intravenous immunoglobulin (IVIg) or plasmapheresis (PE) in part explaining the high mortality and disability compared to treated patients in high-income countries. Added difficulty in traditional PE is its unavailability and specialized device and manpower dependency. Most research in GBS has been conducted in high-income countries, largely in patients with a demyelinating form of GBS. Axonal form of GBS is common in low-income and Asian countries which has a different pathogenesis, clinical course and outcome than the demyelinating form. Very few therapeutic studies have been conducted in low-income countries due to expensive existing modalities of treatment. Here, the investigators propose SVPE as a treatment for GBS in patients from low-income countries. SVPE is relatively cheap, can be done at the bedside without any special device or electricity and eventually is expected to help poor severely affected GBS patients in underdeveloped and developing countries. The main outcomes will be the safety and feasibility of SVPE since this is yet to be established in the resource limited settings. To be able to evaluate the safety of SVPE, additional information will be acquired about the frequency of complications in non-GBS patients with a central line, treated during the same time period at the same study facility as the GBS patients. Severe sepsis due to central line associated blood stream infection and deep venous thrombosis in the limb where the central venous catheter will be inserted during or following the SVPE procedure, will be defined as severe adverse effect (SAE) and will be considered as primary outcome measure for safety. Blood, cerebrospinal fluid and other relevant biological specimens will be analysed for diagnosis and screening for infections. In addition clinical and neurological outcome assessment will be monitored until discharge of the patient from the hospital and up to four weeks since study entry. Confirmation of feasibility and safety, will eventually lead to a randomized control trial in future with a primary focus on the clinical efficacy of SVPE for the treatment of GBS in developing countries as an alternative for the conventional treatment with IVIg or PE.

DETAILED DESCRIPTION:
Study design:

In this safety and feasibility study, 20 GBS patients will be enrolled for SVPE as per protocol criteria. Clinometric measurements (heart rate, blood pressure, temperature, oxygen saturation (SpO2), neurological examination) along with documentation of central line associated blood stream infection (CLABSI) and other complications related to central venous (CV) catheter will be conducted daily and throughout the course of SVPE until the 2nd day of the withdrawal of the CV catheter according to a predefined protocol. Diagnosed or strongly suspected CLABSI and central venous catheter related deep venous thrombosis (DVT) will be followed up for definite outcome to determine the frequency of severe adverse events attributed to CLABSI until the patient discharges from the hospital. Neurological outcome will be documented according to several disability assessment scales throughout the SVPE until discharge and up to four weeks from the enrollment of the GBS patients. In addition, the safety of the SVPE in GBS patients will be compared with the background complication risk by determining the frequency of complications in non-GBS patients treated with a CV catheter at the same intensive care unit (ICU) during the same period using the same protocol for surveillance as in SVPE-treated GBS patients.

SVPE kit:

SVPE kit will be prepared with one blood transfusion set and two saline infusion sets connected with a tri channel device. On the other end the blood transfusion set will be connected with the blood bag, one saline infusion set is connected with 1 liter normal saline mixed with 2500 unit of un fractionated heparin and one saline infusion set is connected with 500 ml hexa-ethyl starch solution. All the tubes should be made air free by fluid column from respective bag. The tri channel is then attached to the central venous catheter.

Procedure of SVPE for GBS patients:

After the SVPE set is prepared, patient's whole blood will be drawn from central venous catheter according to body weight (7 ml/kg) in each session in the blood transfusion bag with gravitation force placing the blood bag below central venous catheter tip level.

The blood column in the transfusion set and in the central venous catheter will be cleared with normal saline mixed heparin solution attached previously through the side channel. The blood bag will be hung beside the patient in a saline stand uninterrupted to separate the plasma and blood cells which will eventually take 2.5 hours with gravitation. Blood cells will be infused back to the patient and plasma will be discarded and replaced by Fresh Frozen Plasma (FFP) and colloid solution alternately in equal volume through the side channel. One blood bag will be used each day for 6 sessions. At the beginning of each session 70 ml of heparin solution will be taken in the blood bag from the heparin mixed normal saline as anticoagulant. Six sessions will be done daily for consecutive 8 days. A total of 48 sessions will be done in eight days. These six sessions of small volume plasma exchange per day in an adult patient will remove approximately 1200 ml of plasma daily and eventually 9600 ml of plasma will be removed in total 48 sessions. All connection ports and tri channels of the central venous catheter, the blood bag and the saline bag are disinfected by using alcohol 70% then dried on air before sampling blood or (dis)connection. These procedures are performed aseptically. Internationally, endorsed guidelines on central venous catheter blood stream infection prevention is followed throughout the entire period of the SVPE procedure. Total active interference with the patient in each session will be 30 minutes and total daily active interference with the patient will be three hours with a Daily schedule at 8AM, 11AM, 2PM, 5PM, 8PM and 11PM. Plasma replacement will be done alternately using fresh frozen plasma and colloid solution (Hexa ethyl starch).

Anticoagulation therapy:

A loading subcutaneous low molecular weight heparin (1.5 mg/kg) will be given at least two hours before the onset of SVPE. Thereafter daily maintenance dose of subcutaneous low molecular weight heparin (1.5 mg/kg) will be continued for eight days or until SVPE completed.

Indication of anti-platelet therapy:

Patients with excessive clotting tendency despite receiving low molecular weight heparin will be subjected for evaluation of platelet activation. If the bleeding time is reduced by >50% of the baseline of the particular GBS patient, investigators will introduce anti-platelet medication. A loading oral dose of aspirin (500 mg) and clopidogrel (600 mg) will be given at least two hours before the next session of SVPE. Thereafter daily maintenance dose of oral aspirin (150 mg) and clopidogrel (75 mg) along with subcutaneous low molecular weight heparin (1.5 mg/kg) will be continued for eight days or until SVPE completed.

Documentation of SVPE procedure:

To define the safety of SVPE, the six daily sessions of SVPE will be documented in terms of duration and amount of the plasma removed in each session, type and volume of replacement fluid and fresh frozen plasma used, and any inconvenience compromising the SVPE sessions temporarily or permanently. Any difficulties hampering SVPE, which currently cannot be anticipated, will be documented as verbatim.

Documentation of hemodynamic parameters and autonomic disturbance:

Throughout the procedure, haemodynamic status including blood pressure, heart rate, any cardiac arrhythmia, oxygen (%) saturation in peripheral blood, fluid intake and output will be monitored daily as per standard practice in all ICU patients. Blood coagulability will be monitored with prothrombin time (PT) and bleeding time (BT) every alternate day. Autonomic parameters will be documented daily as per the presence of high or low blood pressure, increased or decreased pulse rate, orthostatic hypotension, cardiac arrhythmia, bladder and gastrointestinal dysfunction, pupillary abnormality, unusual sweating or hyper salivation.

Documentation of infection:

Features of infections including pyrexia, leukocytosis in peripheral blood, C-reactive protein and evidence of focal infections like positive blood, throat/tracheal aspirate or urine culture for pathogenic organisms etc. will be documented per protocol as per respective standard case record forms for specific hospital acquired infections (HAI). Clinical and laboratory evidence of HAI especially CLABSI will be monitored and explored at anytime during the SVPE procedure until the second day of withdrawal of the central venous catheter. A definite or strongly suspected CLABSI will be followed up until discharge to document the ultimate fate.

Documentation of HAI and complications:

An infection is considered HAI if all elements of a Centers for Disease Control and Prevention/National Healthcare Safety Network (CDC/NHSN) site - specific infection criterion are all present on or after the third calendar day of admission to the facility. Any infection before the third calendar day of admission will be considered as infection present on admission, except in case of CLABSI; which can occur even on day two of central venous catheter insertion. CLABSI, primary and secondary bloodstream infections sepsis and severe sepsis will be the main focus for infection documentation. All the patients eligible as per the enrolment criteria for CLABSI surveillance will be monitored from admission to the ICU. Ventilator associated pneumonia and catheter associated urinary tract infection will also be monitored using established guidelines in order to have a more specific rate of CLABSI and related complications. Appropriate clinical data, imaging, specimens for biochemical and microscopic examination and culture will be documented at specific time points defined as per specific HAI check list . Device associated complications include central venous catheter occlusion, haemorrhage and deep venous thrombosis. All these safety margin indicators will be defined as per specific guideline definitions.

Use antimicrobial agents:

Any infection will be treated by antimicrobial agents accordingly. Choice of the antibiotics (oral or intravenous) will be based on the site of infection, specific organisms isolated and/or severity of the infection reflected in clinical and laboratory features of systemic inflammatory response (raised total white blood cell (WBC) count (>11,000/c mm of blood), C-reactive protein (>40 mg/L) or positive culture of pathogenic organisms) and choices are made after consultation of a microbiologist. Appropriate lower generations of antibiotics for predicted site specific infection will be administered first if necessary before considering subsequent higher generations until the culture sensitivity report is available.

Indications for withholding plasma exchange:

1. Development of severe or terminal concurrent medical illness
2. Hypotension (30 mm Hg decrease of systolic blood pressure or systolic blood pressure<90 or mean arterial pressure (MAP)<65mm Hg) after start of treatment

Indications for resuming plasma exchange:

1. Return of blood pressure to baseline or systolic blood pressure>90 or MAP<65.
2. After management of anaphylactic reaction following FFP or saline infusion.

Indications for replacement of central venous catheter (CVC) to another site:

1. CLABSI or catheter insertion site infection associated with CVC is diagnosed or strongly suspected as per protocol.

Indications for guide wire replacement of central venous catheter (CVC) to the same site:

1. Complete CVC occlusion despite anticoagulant or thrombolytic administration in absence of features of CLABSI

Indication for blood transfusion:

1. Anemia with hemoglobin concentration below 7 gm/dl during and after the SVPE procedure.

When to stop the trial (Stopping rule):

For feasibility purpose: A predictive success rate of 75% will be set regarding the SVPE procedure. If in more than 5 out of 20 SVPE procedure violates the protocol, the procedure will be considered not feasible and modification of the SVPE procedure will be considered before any further re-evaluation of modified procedure for feasibility along with safety.

For safety purpose: A prior distribution of the success rate with regard to severe adverse effect (SAE) will be set as 75%. The investigators will consider severe sepsis due to CLABSI and venous thrombosis related to CVC use as SAE. If >5 patients had SAE at or before completion of SVPE in 20 GBS patients; the study will be stopped. Otherwise an RCT will be planned subsequently to evaluate the neurological efficacy of the SVPE procedure.

Baseline documentation and Initial screening:

Complete blood count including haemoglobin in g/L, total and differential WBC and platelet count and erythrocyte sedimentation rate (ESR), C-reactive protein, prothrombin time, serum creatinine, serum bilirubin and serum glutamic-pyruvic transaminase (SGPT) will be documented as baseline status for GBS patients with SVPE along with screening for hepatitis B, C and HIV.

Documentation of anti-ganglioside antibodies:

Serum concentration of anti-ganglioside antibodies (GM1 and GD1A) will be measured at the beginning and at the end of SVPE to observe the trend in titre change in the serum of GBS patients.

Documentation at the end of SVPE:

On the second day after removal of the central venous line, baseline documentations will be re evaluated. These include complete blood count including haemoglobin in g/L, total and differential WBC and platelet count and ESR, C-reactive protein, prothrombin time, serum creatinine, serum bilirubin and SGPT.

Assessment of neurological function:

Neurological examination will be performed to see the clinical trend of motor, sensory & autonomic parameters before, during the procedure and subsequently in the follow up of the patients up to four weeks.

Assessment of Motor function:

Different clinical assessment scales will be used to monitor changes in motor function. These are the GBS disability Score, Medical Research Council (MRC) sum score, Rasch-built MRC score, Overall Neuropathy Limitation Scale (ONLS), Rasch-built Overall Disability Score (R-ODS).

Sensory function:

Somatic and Gnostic sensation over the limbs will be examined bilaterally. Somatic sensation will be evaluated by examining fine and crud touch and pain sensation over the specific dermatomal regions and gnostic sensation will be evaluated by position & vibration sense.

Autonomic function:

Autonomic parameters will be documented as per the presence of high or low blood pressure, increased or decreased pulse rate, cardiac arrhythmia, bladder and gastrointestinal dysfunction, pupillary abnormality, unusual sweating, hyper salivation and abnormality in hair growth.

ELIGIBILITY:
Inclusion Criteria:

* fulfill the diagnostic criteria for GBS patients of the National Institute of Neurological and Communicative Disorders and Stroke (NINDS) [19]
* ≥ 18 years of age at diagnosis
* unable to walk unaided for more than 10 meters (GBS disability score ≥ 3)
* included within 2 weeks of onset of weakness
* unable to afford standard treatment with IVIg or standard PE
* Informed written consent

Exclusion Criteria:

* previous severe allergic reaction to properly matched blood products
* evidence of healthcare associated infection present on admission (except aspiration pneumonia)
* severe concomitant illness or terminal underlying disease
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-01; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants in whom up to eight liters of plasma could be removed | 8 days
Number of participants who complete forty sessions of SVPE | 8 days
Number of patients developing severe sepsis or septic shock due to CLABSI in SVPE treated GBS patients | 8 days
Number of patients with venous thrombosis in the limb where the central venous catheter | 8 days

SECONDARY OUTCOMES:
Proportion of central venous catheter blockade that requires catheter replacement. | 8 days
Required education time (in days) to acquire expertise to do the SVPE procedure by the responsible staff doctors and nurses | 8 days
Relative risk of CLABSI due to SVPE compared to CLABSI in non-GBS patients treated with a central line at the same ICU | 8 days
Variations of systolic blood pressure greater than 30mm Hg within 30 minutes after starting SVPE | 30 minutes
Proportion of participants in whom SVPE had to be discontinued due to poor hemodynamic tolerance or other side effects and the exact time of discontinuation of the SVPE procedure | 8 days
Development of anaemia (Hb <7 gm./dl) or haemorrhage requiring blood transfusion. | 8 days
Sudden bradycardia involving a reduction of heart rate by more than 20 beats per minute within 30 minutes after starting SVPE | 30 minutes
Rise in heart rate above 120 beats per minute within 30 minutes after starting SVPE | 30 minutes
Improvement by one or more grades in GBS disability score | 4 weeks
  GBS disability score is graded on a scale of 0 - 6
  0: A healthy state
  1. Minor symptoms and capable of running
  2. Able to walk 10 meters or more without assistance but unable to run
  3. Able to walk 10 meters across an open space with help
  4. Bedridden or chair bound
  5. Requiring assisted ventilation for at least part of the day
  6. Dead

CONTACTS AND LOCATIONS:
Overall Officials: Zhahirul Islam, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- National Institute of Neuroscience, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Derived] Islam B, Islam Z, Rahman S, Endtz HP, Vos MC, van der Jagt M, van Doorn PA, Jacobs BC, Mohammad QD. Small volume plasma exchange for Guillain-Barre syndrome in resource-limited settings: a phase II safety and feasibility study. BMJ Open. 2018 Aug 17;8(8):e022862. doi: 10.1136/bmjopen-2018-022862. PMID 30121613
- [Derived] Islam MB, Islam Z, Rahman S, Endtz HP, Vos MC, van der Jagt M, van Doorn PA, Jacobs BC, Mohammad QD. Small volume plasma exchange for Guillain-Barre syndrome in resource poor settings: a safety and feasibility study. Pilot Feasibility Stud. 2017 Sep 29;3:40. doi: 10.1186/s40814-017-0185-0. eCollection 2017. PMID 28975040